CLINICAL TRIAL: NCT02544711
Title: Cost-effectiveness Evaluation of the Use of a Patient Specific Instrument for Surgical Resection of Malignant Bone Tumor Within the Pelvis Versus the Conventional Surgical Treatment
Acronym: MARGIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC15_0097
Record Dates: First submitted 2015-08-24; First posted 2015-09-09 (Estimated); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Sarcoma, Bone Tumor
Keywords: Pelvis; Surgical resection; Patient specific instrument
MeSH Terms: conditions — Sarcoma; Bone Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prospective group :Innovation (Experimental): Surgical treatment using a patient specific instrument (PSI)
  Interventions: Device: Patient specific instrument
- Retrospective group: Reference (Other): Conventional surgical treatment without PSI, using 2D imaging planification
  Interventions: Procedure: Conventional surgical treatment

INTERVENTIONS:
Device: Patient specific instrument — The proposed innovation consists in using patient specific instrument (PSI) for tumor resection. It is compounded of a preoperative assistance to plan the surgery and an intraoperative assistance to reproduce the preoperative planning.
  Other Names: PSI-T; 3D-Side
  Arms: Prospective group :Innovation
Procedure: Conventional surgical treatment — The conventional treatment is planned on two-dimensional images (CT and MRI).
  Arms: Retrospective group: Reference

SUMMARY:
Primitive malignant bone tumor or mixt tumor (compounded of soft tissues and bone) is a rare pathology particularly within the pelvis, the sacrum or the hip (between 25 and 80 new cases in France per year).

The reference treatment is a surgical "en bloc" resection associated or not to a medical treatment. This surgery remains highly challenging because of the complex three-dimensional geometry of the pelvic bone and the proximity of important organs and neurovascular structures. The local recurrence rate is significantly increased when the resection does not respect a safe tissues margin (R0 margin).

A new technology has been developed and used in different reference sites the Patient Specific Instrument (PSI), manufactured by 3D-Side. The PSI allows for a more secure and reliable surgical gesture, leading to more frequent R0 margins.

The main objective of this study is to compare the efficiency of the PSI for bone tumor resections within the pelvis with respect to the reference method.

ELIGIBILITY:
Screening Critieria:

Retrospective group (reference)

* Patient already operated for the same indication as detailed in the prospective group inclusion criteria
* Surgery date within the 6 years before the study activation in the participating center
* Adult (18 years old or more) at the time of surgery

Inclusion Criteria:

Prospective group (innovation)

* Primitive malignant pelvic bone tumor or mixt tumor (primary bone sarcoma, soft tissue sarcoma with bone extension, giant cells tumor of bone and any tumor requiring such a resection)
* Indication for a wide monobloc resection according to clinical guidelines of the pathology ("en bloc" resection of iliac bone including a bone section from periacetabular Enneking zone 2 to the sacrum zone 4, hip extra-articular resection for proximal femur tumors and sacral tumor or ilio-sacral tumors that need a vertical osteotomy or horizontal osteotomy above S2)
* Ability to fill in Euroqol and TESS questionnaires
* Adult (18 years old or more)
* Health insurance holder

Retrospective group (reference)

Patient fulfilling the matching criteria with one patient of the prospective group, according to the following matching criteria (in order of importance):

1. Tumor location (Enneking zones 1, 2, 1-2, 2-3, 1-2-3, 1-2-4, 1-2-3-4, 1-4, sacrum)
2. Tumor type (chondrosarcoma, osteosarcoma, Ewing, chordoma, other tumor type)
3. Surgery center
4. Tumor size (as close as possible between both patients)
5. Response to chemotherapy (good, bad, not applicable).

Exclusion Criteria:

Prospective group (innovation)

* Patient suffering from a local recurrence or a metastasis at recruitment time
* Absence of informed consent
* Pregnancy or breastfeeding
* Minors
* Adults under guardianship or trusteeship

Retrospective group (reference)

* Patient not fulfilling the protocol matching criteria
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2021-05 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
ICER between the innovation treatment group and the reference treatment group. | 3 years
  Incremental Cost-Effectiveness Ratio (ICER) as assessed from the healthcare system perspective: Cost/Local prevented recurrence at 3 years postoperatively

SECONDARY OUTCOMES:
R0, R1 and R2 margin rates | Within 3 years after surgery
  R0, R1 and R2 margin rates as observed by histological exam for each surgical treatment, for each treatment group.
Rate and nature of adverse events related to surgery for each treatment group | Per-operatively and within 3 years after surgery
Quality Of Life (QOL) of patients treated by PSI (prospective group) | 0, 6, 12, 18, 24, 30 and 36 months
  Euroqol questionnaire score
Indirect estimations of means of Quality Adjusted Life Years (QALYs) of patients treated by the reference treatment (retrospective group) extrapolated from QOL of patients treated by PSI (prospective group) | 3 years
  QALYs measures for this group will be extrapolated from the prospective group by estimating the impact of a local recurrence on health-related quality of life.
MSTS score | 12 and 36 months
  Musculoskeletal Tumor Society (MSTS) Score which evaluates 6 items: pain, function, emotional acceptance, walking capacity, technical walking aids, gait.
TESS Score | 12 and 36 months
  Toronto Extremity Salvage Score (TESS) which evaluates 30 items about the global function and patient's activity level.

CONTACTS AND LOCATIONS:
Overall Officials: François Gouin, Professor, Principal Investigator — Nantes University Hospital
Locations (8):
- France (8):
  - Lille University Hospital, Lille
  - Lyon Centre Léon Bérard, Lyon
  - Lyon CRCM Les Massues, Lyon
  - Marseille University Hospital, Marseille
  - Nancy Centre Chirurgical Emile Gallé, Nancy
  - Nantes University Hospital, Nantes
  - Paris Hospital Cochin, Paris
  - Paris Hospital Kremlin-Bicêtre, Paris